CLINICAL TRIAL: NCT02258997
Title: Hepcidin Levels in Sickle Cell Disease (SCD)
Status: Completed | Type: Observational
Sponsor: Kenneth Ataga, MD (Other)
Collaborators: Augusta University (Other)
Responsible Party: Sponsor-Investigator, Kenneth Ataga, MD, Associate Professor of Medicine, Director, University of North Carolina (UNC) Comprehensive Sickle Cell Program, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: 13-2811
Record Dates: First submitted 2014-09-27; First posted 2014-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Sickle Cell Anemia; Sickle - Beta Thalassemia
Keywords: sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HbSS: Subjects are homozygous for the sickle hemoglobin mutation (HbS).
- HbS-beta thalassemia: Subjects are heterozygous for the HbS mutation and beta thalassemia

SUMMARY:
The investigators propose that patients with HbSβ-thalassemia have lower levels of hepcidin and higher levels of GDF-15 than HbSS patients during the non-crisis, "steady states." In addition, the investigators propose that when controlled for RBC transfusion, patients with HbSβ-thalassemia will have higher levels of storage iron (based on serum ferritin).

Participants: Total number of subjects is 42 - 21 subjects with HbSS, and 21 subjects with HbSβ-thalassemia ).

Procedures (methods): Eligible subjects with documented SCD (HbSS, HbS-β 0-thalassemia or HbS-β+-thalassemia) followed at the University of North Carolina (UNC) Comprehensive Sickle Cell Program will be evaluated in this single-center, prospective, cross-sectional study. The patients will be screened for eligibility at the time of a routine sickle cell clinic visit. Patients' data will be obtained in person at the time of evaluation and through review of their medical records. Investigators will obtain information on SCD-related clinical complications and obtain an estimate of the number of lifetime RBC transfusions. Blood samples will be obtained for laboratory tests. Plasma samples for hepcidin, growth differentiation factor 15 (GDF -15), and high-sensitivity CRP will be stored at -80 degrees Celsius until analysis. Other routine laboratory studies including complete blood count (CBC) with differential and reticulocyte count, serum iron profile and ferritin, and liver function tests will be performed at the clinical laboratories of UNC Hospitals.The subjects will have 30 ml. of blood drawn for this research study. Females of child bearing potential will have a urine pregnancy test at the time of the study.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) refers to a group of inherited disorders characterized by the presence of sickle hemoglobin (HbS) that are associated with episodes of acute illness and progressive organ damage. The most common variant of SCD, sickle cell anemia (HbSS), refers to homozygosity for the β S allele, with most of the remaining patients having sickle hemoglobin C disease (HbSC) and sickle beta thalassemia (HbSβ-thalassemia).

SCD may be associated with iron overload that occurs following repeated red blood cell (RBC) transfusions. However, in patients with beta thalassemia major, iron overload occurs due to both repeated RBC transfusions and hyperabsorption of iron. The hyperabsorption of iron in beta thalassemia occurs due to ineffective erythropoiesis and subsequent downregulation of hepcidin. Thalassemia intermedia and major are the most studied human models of hepcidin modulation by ineffective erythropoiesis alone and the combined and opposite effect of both ineffective erythropoiesis and transfusion dependent iron overload, accordingly. Regular transfusions induce massive iron loading but inhibit erythropoietic drive. Accordingly, hepcidin production is higher in thalassemia major than in thalassemia intermedia although still inappropriate to the massive transfusional iron loading that partially counteracts the erythropoietic-dependent hepcidin down-regulation (Origa R et al, 2007; Kattamis A et al, 2006; Camberlein E et al, 2008). No differences in the steady-state levels of hepcidin was observed when HbSS patients (N = 40) were compared with healthy hemoglobin AA (HbAA)controls (N = 30) (85.3 ± 30 l μg/L vs. 83.5 ± 40 l μg/L) (Ezeh C et al, 2005).

Hepcidin is a 25-amino acid peptide produced mainly in the liver and is the major physiological regulator of body iron stores and serum iron. It negatively regulates egress of iron from cells, such as intestinal epithelial cells and macrophages. Growth differentiation factor-15 (GDF-15) and twisted gastrulation protein homolog 1(TWSG1), two transforming growth factor-β (TGF-β) superfamily members released from erythroid precursors, have been proposed to contribute to hepcidin suppression in thalassemia, although it remains unresolved whether GDF-15 and TWSG1 are markers of ineffective erythropoiesis or mediators of hepcidin suppression in vivo.

With the presence of a thalassemia gene, patients with HbSβ-thalassemia (HbSβ0-thalassemia and HbSβ+-thalassemia) may have an increased tendency to absorb excess iron compared to patients with HbSS.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 70 years
* confirmed diagnosis of HbSS or HbS-β thalassemia
* no history of acute vaso-occlusive event (acute pain crisis or acute chest syndrome) requiring emergency room visit or hospitalization over the preceding 4 weeks
* clinically acceptable physical examination and vital signs
* ability of patient or legal representative to understand the requirements of the study and willingness to sign the Informed Consent document.

Exclusion Criteria:

* pregnancy or breastfeeding
* current acute illness, including a painful crisis
* iron deficiency anemia
* history of liver disease with alanine aminotransferase (ALT) ≥ 3 X upper limit of normal (ULN)
* history of hereditary hemochromatosis, connective tissues disease, chronic inflammatory, disorder, or malignancy
* chronic transfusion program or any transfusion within the previous 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the population followed in the Adult Sickle Cell Clinic with either HbSS or HbS-βthalassemia who meet the eligibility criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hepcidin levels in HbSS and HbSβ-thalassemia SCD patients | Assessed at time of enrollment

SECONDARY OUTCOMES:
Levels of GDF-15 in HbSS and HbSβ-thalassemia SCD patients | Assessed at time of enrollment
Ferritin and C-reactive protein (CRP) levels in SCD patients in the non-crisis state | Assessed at time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MBBS, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Background] Origa R, Galanello R, Ganz T, Giagu N, Maccioni L, Faa G, Nemeth E. Liver iron concentrations and urinary hepcidin in beta-thalassemia. Haematologica. 2007 May;92(5):583-8. doi: 10.3324/haematol.10842. PMID 17488680
- [Background] Kattamis A, Papassotiriou I, Palaiologou D, Apostolakou F, Galani A, Ladis V, Sakellaropoulos N, Papanikolaou G. The effects of erythropoetic activity and iron burden on hepcidin expression in patients with thalassemia major. Haematologica. 2006 Jun;91(6):809-12. PMID 16769583
- [Background] Camberlein E, Zanninelli G, Detivaud L, Lizzi AR, Sorrentino F, Vacquer S, Troadec MB, Angelucci E, Abgueguen E, Loreal O, Cianciulli P, Lai ME, Brissot P. Anemia in beta-thalassemia patients targets hepatic hepcidin transcript levels independently of iron metabolism genes controlling hepcidin expression. Haematologica. 2008 Jan;93(1):111-5. doi: 10.3324/haematol.11656. PMID 18166793
- [Background] Ezeh C, Ugochukwu CC, Weinstein J, Okpala I. Hepcidin, haemoglobin and ferritin levels in sickle cell anaemia. Eur J Haematol. 2005 Jan;74(1):86-8. doi: 10.1111/j.1600-0609.2004.00337.x. No abstract available. PMID 15613115